CLINICAL TRIAL: NCT01047436
Title: An Open Label Randomised Comparative Trial to Establish the Efficacy of 3 mg/kg ArTiMist™ When Compared to Intravenous Quinine in Children With Severe or Complicated Falciparum Malaria, or Uncomplicated Falciparum Malaria With Gastrointestinal Complications
Brief Title: Efficacy of ArTiMist™ in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Proto Pharma Ltd (Industry)
Collaborators: Xidea Solutions Limited (Unknown)
Responsible Party: Mr Clive Booles Director of Development, ProtoPharma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART003
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Falciparum Malaria
Keywords: Plasmodium infections; Remittent fever; Artemether; Artemisinins; quinine; Malaria; Protozoan Infections; Anti-Infective Agents; Antiprotozoal Agents; Schistosomicides; Pharmacologic Actions; Malaria, Falciparum; Antimalarials; Antiparasitic Agents; Parasitic Diseases; sublingual
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Protozoan Infections; Parasitic Diseases | interventions — Quinine; Artemether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ArTiMist (artemether sublingual spray) (Experimental)
  Interventions: Drug: Artemether
- Intravenous Quinine (Active Comparator)
  Interventions: Drug: Quinine

INTERVENTIONS:
Drug: Quinine — 20 mg/kg intravenous quinine loading dose, followed by 10 mg/kg intravenously every 8 hours until resumption of normal oral therapy
  Arms: Intravenous Quinine
Drug: Artemether — Artemether sublingual spray 3 mg/kg at protocol specified timepoints until resumption of normal oral therapy
  Other Names: ArTiMist™
  Arms: ArTiMist (artemether sublingual spray)

SUMMARY:
The purpose of this study is to compare the efficacy of Artemether Sublingual Spray (ArTiMist™) with intravenous quinine in children with severe or complicated falciparum malaria, or children with uncomplicated malaria with gastrointestinal complications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's parent or attendant relative has provided informed consent and the patient has assented (where relevant) to participation in the trial
2. The patient is a child that weighs between 5 and 15 kg (kilogram)
3. The patient has falciparum malaria as evidenced by

   1. Thick or thin blood smears of > 500 P falciparum per mcl (microlitre)(patients with mixed infections may be included provided >500 P Falciparum /mcl) and /or
   2. Positive RDT (rapid diagnostic test)for malaria
4. The patient has either

   1. severe or complicated malaria as determined by the Investigator based on the WHO criteria for severity, or
   2. the patient has uncomplicated malaria but is unable to tolerate oral medication as a result of gastrointestinal complications such as vomiting or diarrhoea.

Exclusion Criteria:

1. Attending relative or parent does not provide informed consent for participation, or the child if capable does not assent to participation in the trial.
2. Ability to tolerate oral therapy
3. Patient has received any treatment with an artemisinin or quinine in the last 24 hours
4. Patient has evidence of significant co-infections (this does not include mixed Plasmodium infections).
5. Patient is allergic or intolerant to artemisinins.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, MBChB MBA Dip Pharm Med MFPM, Study Director — Xidea Solutions Limited

REFERENCES:
- [Derived] Bendel D, Rulisa S, Ansah P, Sirima S. Efficacy of a novel sublingual spray formulation of artemether in African children with Plasmodium falciparum malaria. Antimicrob Agents Chemother. 2015 Nov;59(11):6930-8. doi: 10.1128/AAC.00243-15. Epub 2015 Aug 24. PMID 26303805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a single study centre in Rwanda during December 2009.
Groups:
- ArTiMist: Artemether Sublingual Spray 3 mg/kg administered at 0, 8, 24, 36, 48, and 60 hours
- Intravenous Quinine: Intravenous Quinine. Loading dose of 20 mg/kg and subsequent doses of 10 mg/kg 8 hourly
Period: Overall Study
Arm/Group | ArTiMist | Intravenous Quinine
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ArTiMist | Intravenous Quinine | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.03 (1.50) | 3.64 (2.46) | 3.32 (2.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  Rwanda | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Parasitological Success Defined as a Reduction in Parasite Count of ≥ 90% of Baseline at 24 Hours After the First Dose
Time Frame: 24 hours after first dose
Population: For the efficacy endpoints, the analysis was based on the Full Analysis Set (FAS) which was defined as all patients that received at least 1 dose of trial medication and had at least 1 post dose parasite count at 12 h (hours) or 24 h after start of treatment.
Measure: Number; unit: participants
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
participants | 14 | 10
Statistical Analysis 1: Comparison: ArTiMist vs Intravenous Quinine; The sample size was not statistically determined in this initial trial with ArTimist. For the primary outcome analysis, the percentage of patients defined as having success were determined. The difference between ArTiMist and quinine, along with its 95% confidence interval (CI) were determined. The difference between treatments were compared using Fisher's Exact test; Test type: Superiority or Other; p = 0.17, Fisher Exact; difference between treatments = 26.7, 95% CI 2-sided [-0.3 to 53.7]

2. Secondary Outcome: Parasite Clearance Time
Description: Time in hours from the initiation of therapy until the first of two successive parasite-negative smears were obtained
Time Frame: 3h (hours), 6h, 12h, 18h, 24h, 30h, 36h, 48h, 54h, 60h
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
Hours | 35.7 (41.97) | 51.2 (79.04)

3. Primary Outcome: Time for Parasite Count to Fall by 90% PCT(90)
Description: The time taken for the parasite count to fall 90% from baseline
Time Frame: 3h (hours), 6h, 12h, 18h, 24h, 30h, 36h, 48h, 54h, 60h
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
hours | 17.6 (7.34) | 19.8 (13.59)
Statistical Analysis 1: Comparison: ArTiMist vs Intravenous Quinine; The time for the parasite count to fall by 90% (PCT90) was determined for each patient as the time in minutes/seconds, when the parasite count fell by 90% The PCT90 was appropriately summarised for each treatment for the FAS . The times were presented graphically for each endpoint using a life-table curve (Kaplan-Meier method). For each endpoint the survival curves were compared by the log-rank test. The hazard ratio was calculated along with its 95% CI; Test type: Superiority or Other; p = 0.70, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.48 to 3.01]

4. Secondary Outcome: Parasite Reduction Ratio (PRR) at 24 h (Hours) After the First Dose
Description: Reduction in parasitaemia from baseline at 24 h after the first dose of study medication
Time Frame: 24 hours after first dose
Population: For the efficacy endpoints, the analysis was based on the Full Analysis Set (FAS) which was defined as all patients that received at least 1 dose of trial medication and had at least 1 post dose parasite count at 12 h or 24 h
Measure: Median (Full Range); unit: Percent reduction
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
Percent reduction | 100.0 [77 to 100] | 96.9 [53 to 100]

5. Primary Outcome: Time for Parasite Count to Fall by 50% PCT(50)
Description: The time taken for the parasite count to fall 50% from baseline
Time Frame: 3 h (hours) , 6h, 12h, 18h, 24h, 30h, 36h, 48h, 54h, 60h
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
hours | 12.0 (6.48) | 10.8 (7.42)
Statistical Analysis 1: Comparison: ArTiMist vs Intravenous Quinine; The PCT50 was determined for each patient as the time in minutes/seconds, when the parasite count fell by 50% The PCT50 was appropriately summarised for each treatment for the FAS . The times were presented graphically for each endpoint using a life-table curve (Kaplan-Meier method). For each endpoint the survival curves were compared by the log-rank test. The hazard ratio was calculated along with its 95% CI; Test type: Superiority or Other; p = 0.76, Log Rank — Difference between survival curves compared by Log Rank test; Hazard Ratio (HR) = 0.92, 95% CI [0.34 to 2.18]

6. Secondary Outcome: Parasite Reduction Ratio (PRR) at 12 Hours After the First Dose
Description: Reduction in parasitaemia from baseline at 12 hours after the first dose of study medication
Time Frame: 12 h (hours) after first dose
Population: as for outcome 4
Measure: Median (Full Range); unit: Percent reduction
Arm/Group | ArTiMist | Intravenous Quinine
Number analyzed (Participants) | 15 | 15
Percent reduction | 79.6 [-220 to 100] | 75.9 [-58 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the study (01 December 2009) to the last study follow up visit on 19 January 2010
Arm/Group | ArTiMist | Intravenous Quinine
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 13/16 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ArTiMist (N=16) | Intravenous Quinine (N=15)
Malaria reinfection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ArTiMist (N=16) | Intravenous Quinine (N=15)
Anaemia (General disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diarrhoae (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 4 (4)
Pyrexia (General disorders) | 6 (6) | 5 (5)
Bacterial Infection (Infections and infestations) | 0 (0) | 3 (3)
Malaria reinfection (Infections and infestations) | 2 (2) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI was restricted from publishing results for 6 months from the end of the trial. This has now passed and the PI is free to publish the results without restriction